CLINICAL TRIAL: NCT05763225
Title: Validation of the SLEDAI-P/LUPIN Self-questionnaire Completed by the Patient to Measure the Activity of the Systemic Lupus
Brief Title: Validation of Patient E-tool to Measure Systemic Lupus Activity
Acronym: OPTIMISE
Status: Completed | Type: Observational
Sponsor: Association Francaise du Lupus et Autres Maladies Auto-immunes (AFL+) (Other)
Collaborators: Hometrix Health SAS (Other)
Responsible Party: Sponsor
Other Study IDs: nZein
Record Dates: First submitted 2023-02-09; First posted 2023-03-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Patient-reported outcomes; Disease activity; SLEDAI; Patient empowerment; Lupus Erythematosus Systemic; SLEDAI-P; LUPIN
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validation of a self-questionnaire (SLEDAI-P/LUPIN) completed by the patient to measure the activity of the systemic lupus, in order to improve the patient's empowerment.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a rare and chronic autoimmune disease. Disease activity (DA) is marked by remissions, spontaneous relapses or induced by therapeutic modifications. SLE exposes to serious complications requiring close medical follow-up, but flares cannot be predicted and often do not coincide with medical consultations. SLE DA is measured during a consultation using the SLEDAI tool, but cannot be completed by patients. There is therefore high at stake to develop tools allowing patients to measure DA, predict flares and subsequently tailor the medical follow-u to each patient. Using the same framework as a previous nationwide study related to COVID-19 impact (EPICURE survey), we aim to develop and validate, in collaboration with the French national Lupus Reference Centers and Hometrix Health, a patient-tailored tool (SLEDAI-P/LUPIN).

SLEDAI-P/LUPIN was designed by expert lupulogist and patients. It is available as a paper questionnaire and a smartphone app. It consists of simple patient-oriented questions allowing numerical score calculation. In order to validate the SLEDAI-P/LUPIN, we will recruit 500 SLE patients who satisfy the 2019 ACR/EULAR classification criteria. All patients will complete the self-questionnaire and have a follow-up consultation with a clinician within 7 days. The validity of the SLEDAI-P self-questionnaire will be assessed by calculating the correlation between SLEDAI-P/LUPIN and the clinical SLEDAI-2K provided by the clinician (blindly of the SLEDAI-P/LUPIN results). We will also collect information about the quality of life via the SF-36 questionnaire to evaluate if the SLEDAI-P/LUPIN predicts patient-reported outcome measures.

The results of this survey will permit the validation of the SLEDAI-P/LUPIN as a self-questionnaire carried by the patient.

The development of self-administrated disease activity questionnaires such as the SLEDAI-P/LUPIN may allow to better tailor the treatment and follow-up of SLE patients, and empower SLE patients for the control and management of their disease.

ELIGIBILITY:
Inclusion criteria:

Clinical diagnosis of systemic lupus Patient residing in Metropolitan France or in the french Ultra-Marine Departments and Territories Patient who has both completed the SLEDAI-P/LUPIN, SF-12 and been assessed by a specialist via the SLEDAI-2K within 15 days

Exclusion criteria :

Non-lupus patient/participant Patient residing outside France Patient who has not completed the SLEDAI-P/LUPIN OR has not been assessed by a specialist via the SLEDAI-2K within 15 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This survey will be distributed to the entire French population affected by lupus (metropolitan and overseas territories).
  The study is anonymous from the beginning and there will be no way to trace the identity of the participants.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Statistical correlation between the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) questionnaire and the patients reported outcome SLEDAI for Patient / LUpus Patient INdex (SLEDAI-P/LUPIN) | through study completion, an average of 6 months
  Patients reported outcome score versus clinical SLEDAI score, Maximum delay between the two surveys is 7 days. score 0-105 (the highest score represents the highest disease activity)

SECONDARY OUTCOMES:
Quality of life evaluation via the 36-Item Short Form Health Survey (SF-36) | through study completion, an average of 6 months
  The SF-36 has 8 subscales (Physical activity; Limitations due to physical condition; Each of the 8 summary scores is linearly transformed on a scale from 0 (negative to health) to 100 (positive to health)Perceived health; Vitality; Life and relationships with others; Limitations due to psychological condition; Psychological health; Change in perceived health)

CONTACTS AND LOCATIONS:
Locations (31):
- France (29):
  - Médecine interne - Centre hospitalier de la Côte Basque, Bayonne
  - CHU Minjoz, Besançon
  - CHU Bordeaux, Bordeaux
  - Service de Médecine interne et maladies infectieuses (Sud) CHU de Bordeaux-GH Sud - Hôpital Haut-Lévêque, Bordeaux
  - CHU de Clermont-Ferrand - Hôpital Gabriel Montpied Médecine Interne, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - CHU Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - Et service de médecine interne - CHU Réunion site Nord, St Denis, La Réunion
  - Hospices Civils de Lyon, Lyon
  - Hopital de la Croix Rousse - Lyon, Service de médecine Interne, Lyon
  - Médecine Interne - Hôpital Saint Joseph Saint Luc, Lyon
  - Hôpitaux Universitaires de Marseille Conception - Médecine interne, Immunologie et Immunologie clinique, Marseille
  - Service de Médecine Interne de l'Hôpital de la Timone, Marseille
  - Service de médecine interne - Hôpital Nord, Marseille
  - Service de Médecine Interne Hôpital Robert Schuman, Metz
  - CHU de Nancy, Hôpital Brabois, Nancy
  - Service de médecine interne et immunologie clinique CHU de Nancy - Hôpitaux de Brabois, Nancy
  - CHU de Nantes Hôtel Dieu- Centre de compétences maladies systémiques et auto-immunes rares, Nantes
  - Hôpital Saint-Louis - Service de Médecine Interne, Maladies Systémiques, Paris
  - Hôpitaux Universitaires Pitié Salpêtrière - Charles Foix, Paris
  - Hôpital Tenon - Service de dermatologie, médecine vasculaire et allergologie, Paris
  - Hôpital Bicêtre - Service de Rhumatologie, Paris
  - Service de médecine interne CHU de Poitiers, Poitiers
  - Hopital Robert Debre Chu Reims, Reims
  - Département de Médecine Interne du Pr.BENHAMOU CHU DE ROUEN, Rouen
  - Strasbourg University Hospital, Strasbourg
  - Hôpital civil - Immunologie Clinique et Médecine Interne, Strasbourg
  - Service de Médecine Interne & Immunologie Clinique Hôpital Bretonneau CHRU de Tours, Tours
  - CH de Valence - Valence, Service de médecine interne, Valence
- Centre Hospitalier de la Basse Terre, Basse-Terre, Guadeloupe
- Service de Rhumatologie - Médecine Interne 5D CHU de Martinique - Hôpital P. Zobda-Quitman, Martinique, Martinique

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arnaud L, Fagot JP, Mathian A, Paita M, Fagot-Campagna A, Amoura Z. Prevalence and incidence of systemic lupus erythematosus in France: a 2010 nation-wide population-based study. Autoimmun Rev. 2014 Nov;13(11):1082-9. doi: 10.1016/j.autrev.2014.08.034. Epub 2014 Aug 27. PMID 25172239
- [Background] Stoll T, Sutcliffe N, Mach J, Klaghofer R, Isenberg DA. Analysis of the relationship between disease activity and damage in patients with systemic lupus erythematosus--a 5-yr prospective study. Rheumatology (Oxford). 2004 Aug;43(8):1039-44. doi: 10.1093/rheumatology/keh238. Epub 2004 May 25. PMID 15161983
- [Background] Wang C, Mayo NE, Fortin PR. The relationship between health related quality of life and disease activity and damage in systemic lupus erythematosus. J Rheumatol. 2001 Mar;28(3):525-32. PMID 11296953
- [Background] Scherlinger M, Zein N, Gottenberg JE, Riviere M, Kleinmann JF, Sibilia J, Arnaud L. Difficulties and Psychological Impact of the SARS-CoV-2 Pandemic in Patients with Systemic Lupus Erythematosus: A Nationwide Patient Association Study. Healthcare (Basel). 2022 Feb 9;10(2):330. doi: 10.3390/healthcare10020330. PMID 35206945
- [Background] Merrill JT, Neuwelt CM, Wallace DJ, Shanahan JC, Latinis KM, Oates JC, Utset TO, Gordon C, Isenberg DA, Hsieh HJ, Zhang D, Brunetta PG. Efficacy and safety of rituximab in moderately-to-severely active systemic lupus erythematosus: the randomized, double-blind, phase II/III systemic lupus erythematosus evaluation of rituximab trial. Arthritis Rheum. 2010 Jan;62(1):222-33. doi: 10.1002/art.27233. PMID 20039413
- [Background] Stone JH. BLISS! Lupus learns its lessons. Lancet. 2011 Feb 26;377(9767):693-4. doi: 10.1016/S0140-6736(10)61546-2. Epub 2011 Feb 4. No abstract available. PMID 21296404
- [Background] Luijten KM, Tekstra J, Bijlsma JW, Bijl M. The Systemic Lupus Erythematosus Responder Index (SRI); a new SLE disease activity assessment. Autoimmun Rev. 2012 Mar;11(5):326-9. doi: 10.1016/j.autrev.2011.06.011. Epub 2011 Sep 18. PMID 21958603
- [Background] Symmons DP, Coppock JS, Bacon PA, Bresnihan B, Isenberg DA, Maddison P, McHugh N, Snaith ML, Zoma AS. Development and assessment of a computerized index of clinical disease activity in systemic lupus erythematosus. Members of the British Isles Lupus Assessment Group (BILAG). Q J Med. 1988 Nov;69(259):927-37. PMID 3271336
- [Background] Isenberg DA, Garton M, Reichlin MW, Reichlin M. Long-term follow-up of autoantibody profiles in black female lupus patients and clinical comparison with Caucasian and Asian patients. Br J Rheumatol. 1997 Feb;36(2):229-33. doi: 10.1093/rheumatology/36.2.229. PMID 9133936
- [Background] Ravirajan CT, Rowse L, MacGowan JR, Isenberg DA. An analysis of clinical disease activity and nephritis-associated serum autoantibody profiles in patients with systemic lupus erythematosus: a cross-sectional study. Rheumatology (Oxford). 2001 Dec;40(12):1405-12. doi: 10.1093/rheumatology/40.12.1405. PMID 11752513
- [Background] Ehrenstein MR, Conroy SE, Heath J, Latchman DS, Isenberg DA. The occurrence, nature and distribution of flares in a cohort of patients with systemic lupus erythematosus: a rheumatological view. Br J Rheumatol. 1995 Mar;34(3):257-60. doi: 10.1093/rheumatology/34.3.257. PMID 7728402
- [Background] Gordon C, Sutcliffe N, Skan J, Stoll T, Isenberg DA. Definition and treatment of lupus flares measured by the BILAG index. Rheumatology (Oxford). 2003 Nov;42(11):1372-9. doi: 10.1093/rheumatology/keg382. Epub 2003 Jun 16. PMID 12810926
- [Background] Ceccarelli F, Perricone C, Massaro L, Cipriano E, Alessandri C, Spinelli FR, Valesini G, Conti F. Assessment of disease activity in Systemic Lupus Erythematosus: Lights and shadows. Autoimmun Rev. 2015 Jul;14(7):601-8. doi: 10.1016/j.autrev.2015.02.008. Epub 2015 Mar 2. PMID 25742757
- [Background] Isenberg DA, Rahman A, Allen E, Farewell V, Akil M, Bruce IN, D'Cruz D, Griffiths B, Khamashta M, Maddison P, McHugh N, Snaith M, Teh LS, Yee CS, Zoma A, Gordon C. BILAG 2004. Development and initial validation of an updated version of the British Isles Lupus Assessment Group's disease activity index for patients with systemic lupus erythematosus. Rheumatology (Oxford). 2005 Jul;44(7):902-6. doi: 10.1093/rheumatology/keh624. Epub 2005 Apr 6. PMID 15814577
- [Background] Gladman D, Urowitz M, Fortin P, Isenberg D, Goldsmith C, Gordon C, Petri M. Systemic Lupus International Collaborating Clinics conference on assessment of lupus flare and quality of life measures in SLE. Systemic Lupus International Collaborating Clinics Group. J Rheumatol. 1996 Nov;23(11):1953-5. No abstract available. PMID 8923374
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Background] Mosca M, Tani C, Aringer M, Bombardieri S, Boumpas D, Brey R, Cervera R, Doria A, Jayne D, Khamashta MA, Kuhn A, Gordon C, Petri M, Rekvig OP, Schneider M, Sherer Y, Shoenfeld Y, Smolen JS, Talarico R, Tincani A, van Vollenhoven RF, Ward MM, Werth VP, Carmona L. European League Against Rheumatism recommendations for monitoring patients with systemic lupus erythematosus in clinical practice and in observational studies. Ann Rheum Dis. 2010 Jul;69(7):1269-74. doi: 10.1136/ard.2009.117200. Epub 2009 Nov 5. PMID 19892750
- [Background] van Vollenhoven RF, Mosca M, Bertsias G, Isenberg D, Kuhn A, Lerstrom K, Aringer M, Bootsma H, Boumpas D, Bruce IN, Cervera R, Clarke A, Costedoat-Chalumeau N, Czirjak L, Derksen R, Dorner T, Gordon C, Graninger W, Houssiau F, Inanc M, Jacobsen S, Jayne D, Jedryka-Goral A, Levitsky A, Levy R, Mariette X, Morand E, Navarra S, Neumann I, Rahman A, Rovensky J, Smolen J, Vasconcelos C, Voskuyl A, Voss A, Zakharova H, Zoma A, Schneider M. Treat-to-target in systemic lupus erythematosus: recommendations from an international task force. Ann Rheum Dis. 2014 Jun;73(6):958-67. doi: 10.1136/annrheumdis-2013-205139. Epub 2014 Apr 16. PMID 24739325
- [Background] Agmon-Levin N, Mosca M, Petri M, Shoenfeld Y. Systemic lupus erythematosus one disease or many? Autoimmun Rev. 2012 Jun;11(8):593-5. doi: 10.1016/j.autrev.2011.10.020. Epub 2011 Oct 25. PMID 22041578
- [Background] Cervera R, Doria A, Amoura Z, Khamashta M, Schneider M, Guillemin F, Maurel F, Garofano A, Roset M, Perna A, Murray M, Schmitt C, Boucot I. Patterns of systemic lupus erythematosus expression in Europe. Autoimmun Rev. 2014 Jun;13(6):621-9. doi: 10.1016/j.autrev.2013.11.007. Epub 2014 Jan 10. PMID 24418306
- See also: Promoter website — https://lupusplus.com/